CLINICAL TRIAL: NCT06535061
Title: The Effect of White Noise and Pacifier Applications on Pain and Crying Time in Newborns in the Postoperative Period
Brief Title: The Effect of White Noise and Pacifier Applications on Pain and Crying Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Ebru Karaaslan, research assistant, Sanko University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SankoU-Nursing-EK-002
Record Dates: First submitted 2024-07-28; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Newborn
Keywords: White Noise; Pain; Crying Time; Newborn
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: After the newborns left intubation in the postoperative period, physical parameters were measured before, during, after venous blood collection, before, during, after heel blood collection, and before, during and after intravenous intervention, and were evaluated with the Neonatal Infant Pain Scale (NIPS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Pacifiers suitable for the mouth diameter of all newborns were given. Heel blood was collected from the heel of the right foot of all newborns. The heel was stroked by hand before the procedure. Blood flow was accelerated.
  Interventions: Other: white noise
- intervention (Experimental): White noise sound and pacifier implemented Group
  Interventions: Other: white noise

INTERVENTIONS:
Other: white noise — The experimental group was exposed to a white noise sound combined from 4 different sounds: ultrasound heartbeat sound, wave sound, vacuum cleaner sound and hair removal machine sound at 50 dBSPL 5 minutes before the procedure. The experimental group was exposed to white noise for a total of 15 minutes before, during and after the procedure. At the same time, the newborn in the experimental group I was given a pacifier.

SUMMARY:
The objective of the study was to determine the effect of white noise and pacifier applications on pain and crying time in newborns during painful interventions. The research was planned experimentally. Pacifier application was applied to the newborns, who had undergone surgery, and they formed the control group. White noise and pacifier applications were applied to the newborns, who had undergone surgery, and they formed the experimental group.

DETAILED DESCRIPTION:
Data from children's hospitals around the world reveal that pain in pediatric patients from infancy to adolescence is common, under-recognized and undertreated. Compared to adult patients, pediatric patients with the same diagnosis receive fewer doses of analgesics, and the younger children are, the less likely they are to receive adequate analgesia in the medical setting.

A particularly vulnerable group of patients are infants and newborns. During the day, newborns most frequently experience painful interventions such as heel prick blood collection and peripheral venous catheter placement in the neonatal intensive care unit.

Within the scope of the research, no research comparing the effectiveness of white noise and pacifier applications was found in the literature review. By examining this information, the effects of two effective methods on pain management and crying time in newborns in the postoperative period were examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight over 1500 grams
* Having passed the newborn hearing screening test
* Having a history of previous surgery (excluding brain surgeries)
* Not using sedative substances (dormicum, fentanyl)
* Not using opioids
* Having a full stomach 30 minutes before painful interventions
* Having permission from their mothers
* Newborns undergoing blood transfusion only

Exclusion Criteria:

Being intubated

* Having hiberbilirubinemia
* Birth weight below 1500 grams
* Having cerebral palsy
* Having hydrocephalus
* Having spina bifida
* Having had brain surgery

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Neonatal Pain Scale | a day
  The factors evaluated in the neonatal pain scale are facial expression, arms, legs, oxygen saturation, arousal status, breathing pattern, crying, and heart rate factors. It can be preferred in post-operative pain and used for procedural pain. It has 8 parameters in total. A maximum of 7 points can be awarded: 0 points = no pain; 1-2 points = mild pain; 3-4 points = moderate pain; >4 points = severe pain

SECONDARY OUTCOMES:
Neonatal Physiological Evaluation Form | a day
  This form included the newborns' fever, heart rate, respiratory rate and saturation, crying time, and NIPS pain scores 5 minutes before painful interventions, during painful interventions, and 5 minutes after painful interventions. A Nimomed Non-Contact Infrared Thermometer was used to measure the temperature of the newborns. The Nihon Kohden Monitor was used to measure the newborn's heart rate and saturation.
  A newborn scale was used to weigh the newborn's weight. The sound level (lower limit 200-250 Hz, upper limit 10-16 kHz) was evaluated with a Saunal Meter. The newborns were monitored with the above medical instruments. The crying time of the newborns was recorded with a voice recorder, and discussed on a minute basis. The newborn white noise sound was created by combining hair dryer, vacuum cleaner, wave sound and ultrasound device with heartbeat sound. The newborns in the experimental group listened to it for a total of 15 minutes in 5-minute periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Ebru Karaaslan, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided